CLINICAL TRIAL: NCT01043276
Title: A Single Dose, Open, Randomized, 5-Way Crossover Study In Healthy Volunteers To Investigate The Pharmacokinetics Of PF-00258210 Administered Alone Or PF-00258210 Administered Together With PF-00610355 Either As A Free Or A Fixed Dose Combination
Brief Title: A Study To Estimate The Relative Bioavailability Of PF-00258210 Administered Alone Or In Combination With PF-00610355
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B0751001
Record Dates: First submitted 2009-12-07; First posted 2010-01-06 (Estimated); Last update posted 2010-04-27 (Estimated); Status verified 2010-04

CONDITIONS: Asthma
Keywords: Healthy
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Treatment A (Experimental)
  Interventions: Drug: Treatment A
- Treatment B (Experimental)
  Interventions: Drug: Treatment B
- Treatment C (Experimental)
  Interventions: Drug: Treatment C
- Treatment D (Experimental)
  Interventions: Drug: Treatment D
- Treatment E (Experimental)
  Interventions: Drug: Treatment E

INTERVENTIONS:
Drug: Treatment A — PF-00258210 220 µg using inhaler A
  Arms: Treatment A
Drug: Treatment B — PF-00258210 220 µg using inhaler A and 450 µg PF-00610335 using inhaler A
  Arms: Treatment B
Drug: Treatment C — PF-00258210 440 µg and 450 µg PF-00610335 using inhaler A
  Arms: Treatment C
Drug: Treatment D — PF-00258210 350 µg and 450 µg PF-00610335 using inhaler A
  Arms: Treatment D
Drug: Treatment E — PF-00258210 220 µg using inhaler B
  Arms: Treatment E

SUMMARY:
The purpose of this study if to investiagte the time course of PF-00258210 plasma concentration in the presence or absence of PF-00610335 administered via oral inhalation using dry powder inhalers

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 21 and 55 years, inclusive

Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs)

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing)
* A positive urine drug screen
* Pregnant or nursing females

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-01; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
plasma pharmacokinetics AUClast and Cmax | Day 1

SECONDARY OUTCOMES:
plasma pharmacokinetics, AUCinf and Tmax | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0751001&StudyName=A%20Study%20To%20Estimate%20The%20Relative%20Bioavailability%20Of%20PF-00258210%20Administered%20Alone%20Or%20In%20Combination%20With%20PF-00610355